CLINICAL TRIAL: NCT01221818
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single Dose Study of E6007 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E6007-A001-001
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: E6007
- 2 (Experimental)
  Interventions: Drug: E6007
- 3 (Experimental)
  Interventions: Drug: E6007
- 4 (Experimental)
  Interventions: Drug: E6007
- 5 (Experimental)
  Interventions: Drug: E6007
- 6 (Experimental)
  Interventions: Drug: E6007

INTERVENTIONS:
Drug: E6007 — E6007 25mg single dose or matching placebo
  Arms: 1
Drug: E6007 — E6007 50mg single dose or matching placebo
  Arms: 2
Drug: E6007 — E6007 100mg single dose or matching placebo
  Arms: 3
Drug: E6007 — E6007 200mg single dose or matching placebo
  Arms: 4
Drug: E6007 — E6007 400mg single dose or matching placebo
  Arms: 5
Drug: E6007 — E6007 600 mg single dose or matching placebo
  Arms: 6

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single oral ascending doses of E6007 in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, ascending single dose study to evaluate the safety and tolerability of E6007 in healthy subjects. Six dose groups will be evaluated. Subjects will receive either 25 mg, 50 mg, 100 mg, 200 mg, 400 mg, or 600 mg E6007 or matching placebo tablets. Subjects will undergo screening evaluations, baseline evaluations, Day 1 (dosing day), and Days 2-5 evaluations. They will also have a follow-up visit on Day 90 and a Day 180 follow-up phone call.

ELIGIBILITY:
Inclusion criteria:

• Healthy, non-smoking , male or female subjects aged 18-55 years old and with a body mass index (BMI) between 18 and 30 kg/m2 at the time of screening

Exclusion Criteria:

* Evidence of clinically significant infection, hepatic, gastrointestinal, renal, respiratory, endocrine, hematological, neurological, psychiatric, rheumatologic, or musculoskeletal system abnormality based on medical history, physical examination, and screening lab assessments
* History of any gastrointestinal surgery that could impact the absorption of drug
* Evidence of clinically significant cardiovascular abnormality
* Family history of sudden death attributed to cardiac arrhythmia or QTc problems, additional risk factors for torsades de pointes (TdP) (eg, heart failure, hypokalemia, family history of long QT syndrome)
* Known or suspected history of drug or alcohol misuse within 6 months prior to screening, or positive drug or alcohol test
* Positive hepatitis B or C at screening
* Screening laboratory values outside the normal range or have been diagnosed with acquired immune deficiency syndrome (AIDS), or test positive for human immunodeficiency virus (HIV)
* Evidence of clinically significant deviation from normal in physical examination, vital signs, or clinical laboratory assessments at screening
* Known history of any significant drug or food allergy or an ongoing seasonal allergy

  --Known neurological or psychiatric disorder that could impact a neurological assessment
* Known history of autoimmune disease
* History of cancer
* Participated in another clinical trial less than 4 weeks prior to dosing
* Subjects who have received blood products within 4 weeks, donated blood within 8 weeks or donated plasma within 1 week of dosing
* Subjects who have taken dietary supplements (including vitamins), juice, and herbal preparations or other foods or beverage that may affect the various drug metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice and charbroiled meats) within 1 week prior to dosing
* Subjects who used prescription drugs within 4 weeks prior to dosing or over-the-counter (OTC) medications within 1 week prior to dosing
* Subjects who performed strenuous physical activity or exercise within 1 week prior to dosing
* Subjects who answer affirmatively to any of the following questions on the Study Entry Questionnaire: (1) Do you have any medical condition that may make your body unable to fight infections like leukemia, lymphoma, human immunodeficiency virus (HIV), or organ transplant? (2) Over the last 4 weeks have you been treated for cancer and/or for autoimmune diseases; (3) Have you ever taken natalizumab, rituximab, or efalizumab, alemtuzumab, and mycophenolate, or any immunosuppressive agent known to be associated with Progressive Multifocal Leukoencephalopathy (PML)? (4) Have you taken any of the following medicines over the last 12 months: dexamethasone, bethamethasone, methylprednisolone, budesonide, prednisone, methotrexate, cyclosporine, tacrolimus, enbrel, humira, remicade, azathioprine, 6-MP, chemotherapy-related drugs, anti-tumor necrosis factor (TNF) alpha agents, or any immunosuppressive agent other than those associated with Progressive Multifocal Leukoencephalopathy (PML) such as natalizumab, rituximab, efalizumab, alemtuzumab, or mycophenolate?
* Positive John Cunningham Polyomavirus (JCV) blood deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) test result at Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of single oral ascending doses of E6007 in healthy subjects | Day 1 - Day 180

SECONDARY OUTCOMES:
Obtain a preliminary assessment of the pharmacokinetics of these single doses of E6007 | Day 1 - Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Gina Pastino, Study Director — Eisai Inc.
Locations (1):
- Charles River Clinical Services Northwest, Tacoma, Washington, United States